CLINICAL TRIAL: NCT02377596
Title: Assessment of a Feeding Difficulties Diagnostic Tool Questionnaire For Children With Oral Feeding Resistance
Acronym: FDDT
Status: Withdrawn | Type: Observational
Why Stopped: Not enough participants
Sponsor: Benny Kerzner, MD (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Sponsor-Investigator, Benny Kerzner, MD, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: ANUS1108
Record Dates: First submitted 2012-05-14; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Feeding Difficulties; Feeding and Eating Disorders of Childhood
Keywords: Feeding; difficulties; disorders; childhood; eating
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Perceived Feeding Difficulties: To complete the study we will recruit at least 40 of the children perceived by their parents or guardian to have feeding difficulties.

SUMMARY:
Our long term objective is to enhance the pediatrician's management of children with feeding difficulties in a primary care office-based pediatric practice setting. A prerequisite is to rapidly reach an accurate diagnosis so that appropriate therapy can be applied. To improve the efficiency and accuracy of the diagnostic interview the investigators have designed a Feeding Difficulty Diagnostic Tool (FDDT) consisting of a set of questions that fit beneath a 'diagnostic cover' and prompts for basic information. Depending on the answers rendered on the questionnaire particular diagnoses noted on the cover are flagged for consideration.

In this study our specific objectives are 1) to assess the feasibility and acceptability of using the FDDT in the pediatrician's office and 2) to obtain preliminary data on the reliability of using the instrument in the diagnosis and management of children with feeding difficulties.

* Feasibility and acceptability are often interrelated and will be assessed in a broad sense by questionnaires that ascertain, for example, the amount of time needed by parents and staff to fill in and use the FDDT questionnaire, the ease and difficulties encountered in filling out the FDDT questionnaire and the understanding of the questionnaire by the parents.
* Reliability relates to the usefulness of the FDDT questionnaire for the pediatrician in obtaining and organizing the information obtained from the history and physical including anthropometric data to reach a correct diagnosis, the latter being judged in this study against the diagnosis reached independently by trained experts in pediatric feeding difficulties using a modification of their standard diagnostic interview. The frequency of presentation of the various diagnostic sub-categories and the extent of the discrepancy between the conclusions suggested by the FDDT, the pediatrician, and the feeding disorder experts is unknown. Therefore' this pilot study is needed to help determine the sample size necessary to power a more definitive study of the diagnostic tool's accuracy, if necessary. The investigators anticipate that at least three of the categories (children with excessive selectivity, children with demonstrably poor appetite who are vigorous and free of organic disease, and those misperceived to have feeding limitations) will be well represented in this preliminary study.

DETAILED DESCRIPTION:
Background:

Surveys conducted throughout the world repeatedly demonstrate that approximately 50% of mothers consider at least one of their children to have a feeding difficulty, meaning that they resist taking an appropriate amount of food. This implicates between 20% and 30% of all children. The milder cases are frequently considered "picky eaters" and although well nourished they are at significant risk for coercive feeding. This in turn has been associated with cognitive limitations and behavioral problems. Sub-groups do exhibit poor growth, and some have sub-optimal nutrient consumption relative to body size,while others have underlying or co-morbid organic disease. To help identify the relevant intervention for these children, whether it is reassurance for the parents, counseling to resolve behavioral problems (of both the child and the feeder), nutritional intervention and/or medical treatment, it is necessary to identify the separate conditions that contribute to the feeding difficulty and its complications so that appropriate treatment can then be tailored to the cause.

The task of categorizing children with feeding problems is frequently daunting for the pediatrician due to time constraints and lack of training in this field. In developed countries, physicians may refer a child with severe feeding difficulties to a specialist; however, in many parts of the world, these resources are limited or absent. Additionally, health care professionals have a narrow perspective based on their specialized training, whether that is general medical care, specialized care, nutrition, or oral motor therapy.

To overcome the limitations detailed above, a questionnaire was developed based on the work of the principal investigator, Dr. Kerzner and the co-investigator, Dr. Chatoor. This questionnaire is filled out by the parents and their responses prompt the physician to consider relevant diagnostic possibilities for the particular child's feeding difficulty. Once a diagnosis or set of diagnoses is established by utilization of the questionnaire, specific and appropriate therapy can then be provided.

The diagnostic categories that are captured by this tool are based on typical symptoms demonstrated by children with feeding difficulties and their basis has been published by the principal investigator (copy attached).1 Children over one year of age are divided into three groups based on their dominant symptoms: those with poor appetite; those with excessive selectivity; and those with fear of feeding. Children with a poor appetite are further categorized into four sub groups: those who have underlying organic or medical problems; those who are very active and playful but whose poor feeding leads to conflict with the mother; those who fail to-thrive based on poor economic circumstances or neglect; and, finally, those who are eating appropriate amounts of food but are misperceived by their caregivers to have a poor appetite. Each feeding difficulty category has different and unique approaches necessary for its resolution and it is possible for a child to fit into more than one diagnostic category

As the diagnostic nomenclature in the literature has been confusing and in a state of flux there are no data on the relative prevalence of various diagnoses, much less on the diagnostic categories used in the current classification. Consequently, we have minimal guidance for decisions relating to sample size; thus, the need for a pilot study. We believe that this study will allow us an insight into the frequency and variance in diagnosis of at least three of the major categories: children who are vigorous but with poor appetite, those who are highly selective, and those who are in fact misperceived to have a feeding problem. We also have no information on the feasibility and acceptance of the FDDT questionnaire and we believe the pilot study will facilitate our gaining the pediatrician's and office staff's perspective so that in future designs of the instrument we can overcome any practical limitations that become evident.

Design:

This prospective, observational pilot study will be conducted in a single private pediatric office. The pediatricians have incorporated the FDDT questionnaire as a part of the routine evaluation of children coming for "well baby visits". To complete the study we will recruit at least 40 of the children perceived by their parents or guardian to have feeding difficulties. To be sure this number is obtained we will aim to recruit 50 subjects. This study will be approximately one year in duration.

Data Collection:

The following data will be collected on study subjects as illustrated in the flow sheet on page 6 of this research protocol cover sheet.

* Historical data reported by the parent or guardian on the FDDT questionnaire
* The diagnosis suggested on the Cover sheet of the FDDT
* The pediatrician's details of the patient's physical examination, anthropometrics and calculations (weight and length or height percentiles and mid parental height). A prompt for these data is available in the FDDT. The patient's name will blacked out and a study subject number will be inserted.
* Data on the acceptance of the FDDT will be obtained from the office staff, the pediatricians, and the patients' parents.
* The diagnosis reached by the first feeding specialist (CPNP)
* The diagnosis reached by the second feeding specialist (Psychiatrist)

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 12 and 60 months of age
2. Parent or legal guardian is concerned that the patient's feeding behavior is aberrant
3. Parent or legal guardian voluntarily signs and dates an informed consent to participate in the study and provides authorization to use and/or disclose personal health data
4. Parent or legal guardian states their willingness to complete any forms and participate in the telephone interviews needed throughout the study

Exclusion Criteria:

1. Patients with overt, serious organic disease, including:

   * Aspiration with swallowing
   * Developmental delay
   * Cardiorespiratory difficulty interfering with eating
   * Intestinal obstruction
   * Disorders restricting dietary intake, such as diabetes, celiac disease and food allergy f. Known genetic disorders ( e.g., chromosomal trisomies)
2. Patients currently receiving parenteral or supplemental therapeutic enteral nutrition

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This prospective, observational pilot study will be conducted in a single private pediatric office. The pediatricians have incorporated the FDDT questionnaire as a part of the routine evaluation of children coming for "well baby visits". To complete the study we will recruit at least 40 of the children perceived by their parents or guardian to have feeding difficulties. To be sure this number is obtained we will aim to recruit 50 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To determine the degree of concordance between diagnoses arrived at by pediatricians using the FDDT questionnaire with those reached by trained experts in pediatric feeding difficulties using their standard assessment. | during wellness visit (1x) at enrollment
  To determine the degree of concordance between diagnoses arrived at by pediatricians using the FDDT questionnaire (completed in the pediatric office visit) with those reached by trained experts in pediatric feeding difficulties using their standard assessment (completed over the telephone and recorded).
The acceptance and practicality of use of the FDDT by office staff, pediatricians, and patients. (brief questionnaire assessing the practicality of the FDDT measure and the overall acceptance of the measure.) | during wellness visit (1x) at enrollment
  The acceptance and practicality of use of the FDDT by office staff, pediatricians, and patients. The office staff, the pediatricians, and the patients will each fill out a brief questionnaire assessing the practicality of the FDDT measure and the overall acceptance of the measure.

SECONDARY OUTCOMES:
Weight | during wellness visit (1x) at enrollment
  We will collect data on the patient's body weight.
Height | during wellness visit (1x) at enrollment
  We will collect data on the patient's height.
Growth Index | during wellness visit (1x) at enrollment
  We will collect data on the patient's percent of ideal body weight based on weight for height in children less than 2 years of age and body mass index (BMI) in the older child for each of the diagnostic groups

CONTACTS AND LOCATIONS:
Overall Officials: Benny Kerzner, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States